CLINICAL TRIAL: NCT04706611
Title: Efficacy and Safety of Fecal Microbiota Transplantation in Patients With Intestinal Dysbiosis -A Pilot Study
Brief Title: Efficacy and Safety of Fecal Microbiota Transplantation
Acronym: FMT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guangzhou First People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B-2019-041-01
Record Dates: First submitted 2020-12-20; First posted 2021-01-13 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-02

CONDITIONS: Fecal Microbiota Transplantation
MeSH Terms: interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (40):
- Irritable Bowel Syndrome (Experimental): Fecal Microbiota Transplantation will be performed.
  Interventions: Procedure: Fecal Microbiota Transplantation
- Constipation (Experimental): Fecal Microbiota Transplantation will be performed.
  Interventions: Procedure: Fecal Microbiota Transplantation
- Clostridium Difficile Infection (Experimental): Fecal Microbiota Transplantation will be performed.
  Interventions: Procedure: Fecal Microbiota Transplantation
- Functional Dyspepsia (Experimental): Fecal Microbiota Transplantation will be performed.
  Interventions: Procedure: Fecal Microbiota Transplantation
- Parkinson's Disease (Experimental): Fecal Microbiota Transplantation will be performed.
  Interventions: Procedure: Fecal Microbiota Transplantation
- Metabolic Syndrome (Experimental): Fecal Microbiota Transplantation will be performed.
  Interventions: Procedure: Fecal Microbiota Transplantation
- Non-Alcoholic Fatty Liver Disease (Experimental): Fecal Microbiota Transplantation will be performed.
  Interventions: Procedure: Fecal Microbiota Transplantation
- Autism Spectrum Disorder (Experimental): Fecal Microbiota Transplantation will be performed.
  Interventions: Procedure: Fecal Microbiota Transplantation
- Radiation Enteritis (Experimental): Fecal Microbiota Transplantation will be performed.
  Interventions: Procedure: Fecal Microbiota Transplantation
- Atopic Dermatitis (Experimental): Fecal Microbiota Transplantation will be performed.
  Interventions: Procedure: Fecal Microbiota Transplantation
- Food Allergic (Experimental): Fecal Microbiota Transplantation will be performed.
  Interventions: Procedure: Fecal Microbiota Transplantation
- Graft-versus-Host Disease (Experimental): Fecal Microbiota Transplantation will be performed.
  Interventions: Procedure: Fecal Microbiota Transplantation
- Obesity (Experimental): Fecal Microbiota Transplantation will be performed.
  Interventions: Procedure: Fecal Microbiota Transplantation
- Diabetes mellitus (Experimental): Fecal Microbiota Transplantation will be performed.
  Interventions: Procedure: Fecal Microbiota Transplantation
- Multi-Drug Resistant Infection (Experimental): Fecal Microbiota Transplantation will be performed.
  Interventions: Procedure: Fecal Microbiota Transplantation
- Hepatic Encephalopathy (Experimental): Fecal Microbiota Transplantation will be performed.
  Interventions: Procedure: Fecal Microbiota Transplantation
- Enteric Dysbacteriosis (Experimental): Fecal Microbiota Transplantation will be performed.
  Interventions: Procedure: Fecal Microbiota Transplantation
- Multiple Sclerosis (Experimental): Fecal Microbiota Transplantation will be performed.
  Interventions: Procedure: Fecal Microbiota Transplantation
- Pseudomembranous Enteritis (Experimental): Fecal Microbiota Transplantation will be performed.
  Interventions: Procedure: Fecal Microbiota Transplantation
- Acute Pancreatitis (Experimental): Fecal Microbiota Transplantation will be performed.
  Interventions: Procedure: Fecal Microbiota Transplantation
- Chronic Fatigue Syndrome (Experimental): Fecal Microbiota Transplantation will be performed.
  Interventions: Procedure: Fecal Microbiota Transplantation
- Acute-on-chronic Liver Failure with HBV Infection (Experimental): Fecal Microbiota Transplantation will be performed.
  Interventions: Procedure: Fecal Microbiota Transplantation
- Alcoholic Liver Disease (Experimental): Fecal Microbiota Transplantation will be performed.
  Interventions: Procedure: Fecal Microbiota Transplantation
- Anorexia (Experimental): Fecal Microbiota Transplantation will be performed.
  Interventions: Procedure: Fecal Microbiota Transplantation
- Decompensated Cirrhosis (Experimental): Fecal Microbiota Transplantation will be performed.
  Interventions: Procedure: Fecal Microbiota Transplantation
- Henoch-Schonlein Purpura (Experimental): Fecal Microbiota Transplantation will be performed.
  Interventions: Procedure: Fecal Microbiota Transplantation
- Autoimmune Liver Disease (Experimental): Fecal Microbiota Transplantation will be performed.
  Interventions: Procedure: Fecal Microbiota Transplantation
- Systemic Lupus Erythematosus (Experimental): Fecal Microbiota Transplantation will be performed.
  Interventions: Procedure: Fecal Microbiota Transplantation
- IgG4-Related Disease (Experimental): Fecal Microbiota Transplantation will be performed.
  Interventions: Procedure: Fecal Microbiota Transplantation
- Celiac Disease (Experimental): Fecal Microbiota Transplantation will be performed.
  Interventions: Procedure: Fecal Microbiota Transplantation
- Protein-losing Enteropathy (Experimental): Fecal Microbiota Transplantation will be performed.
  Interventions: Procedure: Fecal Microbiota Transplantation
- Asperger Syndrome (Experimental): Fecal Microbiota Transplantation will be performed.
  Interventions: Procedure: Fecal Microbiota Transplantation
- Rheumatoid arthritis (Experimental): Fecal Microbiota Transplantation will be performed.
  Interventions: Procedure: Fecal Microbiota Transplantation
- Ulcerative colitis (Experimental): Fecal Microbiota Transplantation will be performed.
  Interventions: Procedure: Fecal Microbiota Transplantation
- Crohn's disease (Experimental): Fecal Microbiota Transplantation will be performed.
  Interventions: Procedure: Fecal Microbiota Transplantation
- Psoriasis (Experimental): Fecal Microbiota Transplantation will be performed.
  Interventions: Procedure: Fecal Microbiota Transplantation
- Ankylosing spondylitis (Experimental): Fecal Microbiota Transplantation will be performed.
  Interventions: Procedure: Fecal Microbiota Transplantation
- Immune checkpoint inhibition-related colitis (Experimental): Fecal Microbiota Transplantation will be performed.
  Interventions: Procedure: Fecal Microbiota Transplantation
- Autoimmune enteropathy (Experimental): Fecal Microbiota Transplantation will be performed.
  Interventions: Procedure: Fecal Microbiota Transplantation
- Drug-induced diarrhea (Experimental): Fecal Microbiota Transplantation will be performed.
  Interventions: Procedure: Fecal Microbiota Transplantation

INTERVENTIONS:
Procedure: Fecal Microbiota Transplantation — Procedure: Fecal Microbiota Transplantation

SUMMARY:
In recent years, researches illustrate that multifactorial diseases such as functional gastrointestinal disorders, autoimmune diseases, metabolic, behavioral and neurological diseases are associated with an abnormal microbiome structure-dysbiosis, which means the imbalance of the microbiome community. Fecal microbiota transplantation (FMT), the infusion of faeces from a healthy donor to the gastrointestinal tract of a recipient patient aiming to alter the intestine microbiota, is recommended to be performed in Clostridium difficile infection(CDI) as the most effective therapy. It also being used experimentally in the treatment of the disease states linked to dysbiosis of the intestinal microbiota. However, the efficacy and safety of FMT to treat the dysbiosis-associated diseases is still in its infancy. To further verify the indications above, more data is required to be collected through studies.

ELIGIBILITY:
Inclusion Criteria:

Confirmed diagnosis of any of following diseases:

* Irritable Bowel Syndrome
* Ulcerative colitis
* Crohn's disease
* Constipation
* Clostridium Difficile Infection
* Functional Dyspepsia
* Parkinson's Disease
* Metabolic Syndrome
* Non-Alcoholic Fatty Liver Disease
* Autism Spectrum Disorder
* Radiation Enteritis
* Atopic Dermatitis
* Food Allergic
* Graft-versus-Host Disease
* Obesity
* Diabetes mellitus
* Multi-Drug Resistant Infection
* Hepatic Encephalopathy
* Enteric Dysbacteriosis
* Multiple Sclerosis
* Pseudomembranous Enteritis
* Acute Pancreatitis
* Chronic Fatigue Syndrome
* Acute-on-chronic Liver Failure with HBV Infection
* Alcoholic Liver Disease
* Anorexia
* Decompensated Cirrhosis
* Henoch-Schonlein Purpura
* Autoimmune Liver Disease
* Systemic Lupus Erythematosus
* Rheumatoid arthritis
* IgG4-Related Disease
* Celiac Disease
* Protein-losing Enteropathy
* Asperger Syndrome
* Rheumatoid arthritis
* Psoriasis
* Ankylosing spondylitis
* Immune checkpoint inhibition-related colitis
* Autoimmune enteropathy
* Drug-induced diarrhea
* Suffering from gastrointestinal symptoms such as constipation, diarrheas, abdominal pain, flatulence, etc.
* The participants must be able to tolerate the FMT infusion method such as endoscopy, colonoscopy, capsule, nasoduodenal tube insertion, etc.

Exclusion Criteria:

* Current pregnancy or breast-feeding;
* Suffering from other severe diseases, including liver or kidney failure, heart failure, MODS, coma, cerebrovascular accident;
* Known contraindication to all FMT infusion method such as nasoduodenal tube insertion, endoscopy, colonoscopy and enema;
* Any conditions that may render the efficacy of FMT or at the discretion of the investigators.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-01-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The efficacy of FMT in patients with gastrointestinal symptom will be assessed by the change of Gastrointestinal Symptom Rating Scale(GSRS). | 1 year
  Gastrointestinal Symptom Rating Scale(GSRS) is a measure of gastrointestinal symptom severity in five clusters (pain, bloating, constipation, diarrhea, and early satiety).The items are scored between 1 and 7, where 1 corresponds to "no discomfort at all" and 7 to "very severe discomfort" from the symptom. The participants will be asked to filled in the scale in several time points from baseline to 12 months after FMT.

SECONDARY OUTCOMES:
Number of Participants With Treatment-Related Adverse Events as Assessed by Common Terminology Criteria for Adverse Events(CTCAE) V4.0 | 1 year

OTHER OUTCOMES:
Numbers of patients who have improvement in clinical symptoms (depends on each disease as stated in outcome) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Hongli Huang, MM, Principal Investigator — Guangzhou First People's Hospital
Locations (1):
- Guangzhou First People's Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Levy M, Kolodziejczyk AA, Thaiss CA, Elinav E. Dysbiosis and the immune system. Nat Rev Immunol. 2017 Apr;17(4):219-232. doi: 10.1038/nri.2017.7. Epub 2017 Mar 6. PMID 28260787
- [Background] Brandt LJ. American Journal of Gastroenterology Lecture: Intestinal microbiota and the role of fecal microbiota transplant (FMT) in treatment of C. difficile infection. Am J Gastroenterol. 2013 Feb;108(2):177-85. doi: 10.1038/ajg.2012.450. Epub 2013 Jan 15. PMID 23318479
- [Background] Paramsothy S, Kamm MA, Kaakoush NO, Walsh AJ, van den Bogaerde J, Samuel D, Leong RWL, Connor S, Ng W, Paramsothy R, Xuan W, Lin E, Mitchell HM, Borody TJ. Multidonor intensive faecal microbiota transplantation for active ulcerative colitis: a randomised placebo-controlled trial. Lancet. 2017 Mar 25;389(10075):1218-1228. doi: 10.1016/S0140-6736(17)30182-4. Epub 2017 Feb 15. PMID 28214091
- [Background] Ooijevaar RE, Terveer EM, Verspaget HW, Kuijper EJ, Keller JJ. Clinical Application and Potential of Fecal Microbiota Transplantation. Annu Rev Med. 2019 Jan 27;70:335-351. doi: 10.1146/annurev-med-111717-122956. Epub 2018 Nov 7. PMID 30403550
- [Background] Lee P, Yacyshyn BR, Yacyshyn MB. Gut microbiota and obesity: An opportunity to alter obesity through faecal microbiota transplant (FMT). Diabetes Obes Metab. 2019 Mar;21(3):479-490. doi: 10.1111/dom.13561. Epub 2018 Nov 20. PMID 30328245
- [Background] Bajaj JS, Kassam Z, Fagan A, Gavis EA, Liu E, Cox IJ, Kheradman R, Heuman D, Wang J, Gurry T, Williams R, Sikaroodi M, Fuchs M, Alm E, John B, Thacker LR, Riva A, Smith M, Taylor-Robinson SD, Gillevet PM. Fecal microbiota transplant from a rational stool donor improves hepatic encephalopathy: A randomized clinical trial. Hepatology. 2017 Dec;66(6):1727-1738. doi: 10.1002/hep.29306. Epub 2017 Oct 30. PMID 28586116
- [Background] Sun MF, Zhu YL, Zhou ZL, Jia XB, Xu YD, Yang Q, Cui C, Shen YQ. Neuroprotective effects of fecal microbiota transplantation on MPTP-induced Parkinson's disease mice: Gut microbiota, glial reaction and TLR4/TNF-alpha signaling pathway. Brain Behav Immun. 2018 May;70:48-60. doi: 10.1016/j.bbi.2018.02.005. Epub 2018 Feb 20. PMID 29471030
- [Background] Johnsen PH, Hilpusch F, Cavanagh JP, Leikanger IS, Kolstad C, Valle PC, Goll R. Faecal microbiota transplantation versus placebo for moderate-to-severe irritable bowel syndrome: a double-blind, randomised, placebo-controlled, parallel-group, single-centre trial. Lancet Gastroenterol Hepatol. 2018 Jan;3(1):17-24. doi: 10.1016/S2468-1253(17)30338-2. Epub 2017 Nov 1. PMID 29100842
- [Background] El-Salhy M, Hatlebakk JG, Gilja OH, Brathen Kristoffersen A, Hausken T. Efficacy of faecal microbiota transplantation for patients with irritable bowel syndrome in a randomised, double-blind, placebo-controlled study. Gut. 2020 May;69(5):859-867. doi: 10.1136/gutjnl-2019-319630. Epub 2019 Dec 18. PMID 31852769
- [Background] Leshem A, Horesh N, Elinav E. Fecal Microbial Transplantation and Its Potential Application in Cardiometabolic Syndrome. Front Immunol. 2019 Jun 14;10:1341. doi: 10.3389/fimmu.2019.01341. eCollection 2019. PMID 31258528
- [Background] DeFilipp Z, Bloom PP, Torres Soto M, Mansour MK, Sater MRA, Huntley MH, Turbett S, Chung RT, Chen YB, Hohmann EL. Drug-Resistant E. coli Bacteremia Transmitted by Fecal Microbiota Transplant. N Engl J Med. 2019 Nov 21;381(21):2043-2050. doi: 10.1056/NEJMoa1910437. Epub 2019 Oct 30. PMID 31665575